CLINICAL TRIAL: NCT02377128
Title: Ovarian Reserve Following Bilateral Salpingectomy Versus Tubal Ligation During Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Hadas Ganer Herman, Dr., Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0028-15-WOMC
Record Dates: First submitted 2015-02-15; First posted 2015-03-03 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Ovarian Reserve
Keywords: Study; focus; ovarian; reserve
MeSH Terms: interventions — Sterilization, Tubal

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Bilateral salpingectomy (Experimental): Cesarean section with bilateral salpingectomy
  Interventions: Procedure: Bilateral salpingectomy
- Tubal ligation (Active Comparator): Cesarean section with tubal ligation
  Interventions: Procedure: Tubal ligation
- No intervention (No Intervention): Cesarean section with no additional intervention

INTERVENTIONS:
Procedure: Bilateral salpingectomy — Surgical bilateral removal of fallopian tubes (not involving ovaries)
  Arms: Bilateral salpingectomy
Procedure: Tubal ligation — Bilateral ligation of fallopian tubes (not involving ovaries)
  Arms: Tubal ligation

SUMMARY:
The aforementioned study was designed to evaluate short term ovarian reserve as assessed by anti-Mullerian hormone(AMH) levels following bilateral salpingectomy versus tubal ligation, as part of cesarean sections performed in women requesting future sterilization. The investigators aim to recruit 3 groups of 15 women undergoing elective cesarean section at the investigators' institution, 2 of which request sterilization (allocated to tubal ligation or bilateral salpingectomy) and one undergoing solely cesarean section. The groups will have blood drawn for AMH prior to the procedure and at a post-operation visit 8 weeks following. This is preformed in light of validated data offering better sterilization and possible diminished future risk of ovarian cancer with salpingectomy. Also, is has been proved to be just as safe as tubal ligation. This will be performed as a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing elective cesrean section at the investigators' institution, requesting sterilization, willing to have blood withdrawn for AMH levels prior to surgery, willing to participate in 8 weeks post-operation follow up with blood withdrawn

Exclusion Criteria:

* Non-elective cesarean section, non willing to have blood withdrawn or participate in follow up, prior salpingectomy, prior premature ovarian failure/egg donation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Anti Mullerian hormone (AMH) levels ng/mL at 8 weeks | Baseline and 8 weeks following surgery
  AMH levels

REFERENCES:
- [Background] McAlpine JN, Hanley GE, Woo MM, Tone AA, Rozenberg N, Swenerton KD, Gilks CB, Finlayson SJ, Huntsman DG, Miller DM; Ovarian Cancer Research Program of British Columbia. Opportunistic salpingectomy: uptake, risks, and complications of a regional initiative for ovarian cancer prevention. Am J Obstet Gynecol. 2014 May;210(5):471.e1-11. doi: 10.1016/j.ajog.2014.01.003. Epub 2014 Jan 9. PMID 24412119
- [Background] Erickson BK, Conner MG, Landen CN Jr. The role of the fallopian tube in the origin of ovarian cancer. Am J Obstet Gynecol. 2013 Nov;209(5):409-14. doi: 10.1016/j.ajog.2013.04.019. Epub 2013 Apr 10. PMID 23583217
- [Background] Kamran MW, Vaughan D, Crosby D, Wahab NA, Saadeh FA, Gleeson N. Opportunistic and interventional salpingectomy in women at risk: a strategy for preventing pelvic serous cancer (PSC). Eur J Obstet Gynecol Reprod Biol. 2013 Sep;170(1):251-4. doi: 10.1016/j.ejogrb.2013.06.030. Epub 2013 Jul 21. PMID 23880597
- [Background] Rosenblatt KA, Thomas DB. Reduced risk of ovarian cancer in women with a tubal ligation or hysterectomy. The World Health Organization Collaborative Study of Neoplasia and Steroid Contraceptives. Cancer Epidemiol Biomarkers Prev. 1996 Nov;5(11):933-5. PMID 8922304
- [Background] Falconer H, Yin L, Gronberg H, Altman D. Ovarian cancer risk after salpingectomy: a nationwide population-based study. J Natl Cancer Inst. 2015 Jan 27;107(2):dju410. doi: 10.1093/jnci/dju410. Print 2015 Feb. PMID 25628372
- [Background] Committee opinion no. 620: Salpingectomy for ovarian cancer prevention. Obstet Gynecol. 2015 Jan;125(1):279-281. doi: 10.1097/01.AOG.0000459871.88564.09. PMID 25560145
- [Background] Ghezzi F, Cromi A, Siesto G, Bergamini V, Zefiro F, Bolis P. Infectious morbidity after total laparoscopic hysterectomy: does concomitant salpingectomy make a difference? BJOG. 2009 Mar;116(4):589-93. doi: 10.1111/j.1471-0528.2008.02085.x. PMID 19250369
- [Background] Sezik M, Ozkaya O, Demir F, Sezik HT, Kaya H. Total salpingectomy during abdominal hysterectomy: effects on ovarian reserve and ovarian stromal blood flow. J Obstet Gynaecol Res. 2007 Dec;33(6):863-9. doi: 10.1111/j.1447-0756.2007.00669.x. PMID 18001455
- [Background] Morelli M, Venturella R, Mocciaro R, Di Cello A, Rania E, Lico D, D'Alessandro P, Zullo F. Prophylactic salpingectomy in premenopausal low-risk women for ovarian cancer: primum non nocere. Gynecol Oncol. 2013 Jun;129(3):448-51. doi: 10.1016/j.ygyno.2013.03.023. Epub 2013 Apr 2. PMID 23558052
- [Background] Findley AD, Siedhoff MT, Hobbs KA, Steege JF, Carey ET, McCall CA, Steiner AZ. Short-term effects of salpingectomy during laparoscopic hysterectomy on ovarian reserve: a pilot randomized controlled trial. Fertil Steril. 2013 Dec;100(6):1704-8. doi: 10.1016/j.fertnstert.2013.07.1997. Epub 2013 Aug 29. PMID 23993887
- [Background] Peterson HB, Xia Z, Hughes JM, Wilcox LS, Tylor LR, Trussell J. The risk of ectopic pregnancy after tubal sterilization. U.S. Collaborative Review of Sterilization Working Group. N Engl J Med. 1997 Mar 13;336(11):762-7. doi: 10.1056/NEJM199703133361104. PMID 9052654
- [Result] Koninger A, Kauth A, Schmidt B, Schmidt M, Yerlikaya G, Kasimir-Bauer S, Kimmig R, Birdir C. Anti-Mullerian-hormone levels during pregnancy and postpartum. Reprod Biol Endocrinol. 2013 Jul 11;11:60. doi: 10.1186/1477-7827-11-60. PMID 23844593
- [Result] La Marca A, Giulini S, Orvieto R, De Leo V, Volpe A. Anti-Mullerian hormone concentrations in maternal serum during pregnancy. Hum Reprod. 2005 Jun;20(6):1569-72. doi: 10.1093/humrep/deh819. Epub 2005 Feb 25. PMID 15734752
- [Derived] Ganer Herman H, Gluck O, Keidar R, Kerner R, Kovo M, Levran D, Bar J, Sagiv R. Ovarian reserve following cesarean section with salpingectomy vs tubal ligation: a randomized trial. Am J Obstet Gynecol. 2017 Oct;217(4):472.e1-472.e6. doi: 10.1016/j.ajog.2017.04.028. Epub 2017 Apr 25. PMID 28455082